CLINICAL TRIAL: NCT04113213
Title: Primary Care - Prescribing Lifestyle Adjustments for Cardiovascular Health (Phase II)
Brief Title: Primary Care - Prescribing Lifestyle Adjustments for Cardiovascular Health
Acronym: P-PLAC 2
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: CV-19 pandemic
Sponsor: University of South Wales (Other)
Collaborators: Public Health Wales (Other Government); Cwm Taf University Health Board (NHS) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 260480
Record Dates: First submitted 2019-07-19; First posted 2019-10-02 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Behavior Change Interventions; Cardiovascular Diseases; Cardiovascular Risk Factor; Behavior, Health
MeSH Terms: conditions — Cardiovascular Diseases; Health Behavior

STUDY DESIGN:
Intervention Model Description: The study is an interventional controlled observational study based in the Primary Care setting. Control groups will be utilized through the mechanism of wait-listing the enrolment of recruitment centres into the study.
  Mixed methods will be used for both data collection and analysis. Historical clinical participant data (pre-intervention - from 12months) will be collected by the PI. Data will be collected immediately after the consultation and at 3 months post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard care during consultations.
- Intervention (Experimental): Standard care during consultations with the addition of a physical lifestyle prescription.
  Interventions: Behavioral: Lifestyle Prescription (LRx)

INTERVENTIONS:
Behavioral: Lifestyle Prescription (LRx) — Lifestyle prescription, based on the UK WP10 medicinal prescription form. Includes advice and guidance regarding physical activity, diet, smoking and alcohol consumption.
  Arms: Intervention

SUMMARY:
Prescribing lifestyle changes to patients who are at risk of cardiovascular disease, may be an extremely cost effective mechanism of improving health for the individual themselves and the NHS. It is already proven that positive lifestyle changes such as improved diet, increased physical activity, quitting smoking and reducing alcohol consumption can lower the risk of cardiovascular disease, as well as reduce the risk of all-cause mortality.

P-PLAC2 (Primary Care - Prescribing Lifestyle Adjustments for Cardiovascular Health) is a Phase II interventional study to determine the efficacy of a Lifestyle Prescription (LRx), from the viewpoint of patients and healthcare practitioners. The study uses a mixed methods design, and full study training and support will be provided to staff involved in the recruitment of patients, through to the behaviour change consultation, and end of study.

If the study proves successful, a lifestyle prescription (LRx) could then be made available to support NHS staff throughout all disciplines (specifically those working with patients who are at risk of cardiovascular disease (CVD).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over.
* Able and willing to provide written informed consent.
* Understands spoken and written English.

Exclusion Criteria:

* Participant is unwilling or unable to provide written informed consent.
* Participant is pregnant.
* Participant has a diagnosed psychological disorder.
* Participant has a drug dependency.
* Participant is housebound, or resides in a nursing home.
* Participant has behavioural issues or learning difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-10-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
A prescription (LRx) being issued during a consultation | During month 7 of the study
  Number of a co- signed prescription (LRx) forms. Total number of forms to be co-signed = 120.
Patient view of the prescription (LRx) and consultation Questionnaire | During month 7 of the study
  Completed study questionnaires. Total number of questionnaires to be completed = 120. Responses will be recorded to gain feedback from the patient participants regarding their thoughts and feelings of their consultation with and without the intervention of the prescription (LRx) - control vs interventional group. Initials responses from the questionnaires will be compared with the participants 3mth post consultation questionnaire to establish if they acted upon the guidance offered, and if they're thought and feelings had changed during the time.
  Scale: 7 (minimum) to 41 (maximum). A lower value represents a better (more positive) outcome.
Healthcare Practitioner (HCP) view of the prescription (LRx) and consultation Questionnaire | during month 7 of the study
  Completed clinician questionnaires. Total number of questionnaires to be completed = 12. Responses will be recorded to gain feedback from the clinicians regarding their thoughts and feelings of their consultations with and without the intervention of the prescription (LRx).
  Sections 1 to 3:
  Section 1 Scale: 9 to 54 (a lower score represents a better, more positive outcome) Section 2 Scale: 8 to 48 (a lower score represents a better, more positive outcome) Section 3 Scale: 6 to 36 (a lower score represents a better, more positive outcome)
  Total score available: 23 to 138

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Wales, Pontypridd, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No